CLINICAL TRIAL: NCT06126432
Title: National Cheng Kung University Hospital
Brief Title: Beneficial Effects of Probiotics on Improvement of Gut Dysbiosis and Ascending Cholangitis in Patients Received Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-ER-103-318
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Precancerous Lesions
Keywords: Ampullary; Pancreas

STUDY DESIGN:
Intervention Model Description: Single intervention arm with trial treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To evaluate the effects of probiotics consumption (Experimental): Subjects consumed 2 bottles of probiotics-containing yogurt per day for 1 month
  Interventions: Dietary Supplement: Yugart

INTERVENTIONS:
Dietary Supplement: Yugart — Yugart 2 bottles per day for 1 month

SUMMARY:
To determine whether probiotics have beneficial effect on gut dysbiosis and postoperative ascending cholangitis in patients with pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Gut dysbiosis and postoperative ascending cholangitis (POAC) occurred after pancreaticoduodenectomy (PD). To date, no clinical trial has evaluated the association between gut dysbiosis, POAC and probiotics. POAC is a common morbidity after pancreaticoduodenectomy or in obstructive jaundice patients with endoscopic retrograde biliary drainage (ERBD). It frequently induces longer hospital stay and makes the major obstacle for postoperative chemotherapy. This phenomenon reveals the important role of ampullary vater in control of retrograde bacterial inflow into bile duct. However, the exact difference of gut microbiota after pancreaticoduodenectomy is still unknown. Probiotics is reported efficacy in restore the normal flora of gut microbiota. So, this study is to evaluate the effects of probiotics consumption, Yugart 2 bottles per day for 1 month on gut microbiota in control of ascending cholangitis before and after pancreaticoduodenectomy through the analysis of microbial community by next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with peri-ampullary lesions and scheduled to receive pancreaticoduodenectomy (PD) were designed as experimental group; subjects with pancreatic lesions and scheduled to receive distal pancreatectomy (DP) were designed as control group.
* Subjects that already received PD for more than 6 months to join the study and aim to evaluate the effect of probiotics on gut microbiota and postoperative ascending cholangitis (POAC).
* Subjects with the amount of two bottles a day (one provided in the morning and the other in the afternoon) for a duration of 4 weeks.

Exclusion Criteria:

* Subjects are currently participating in any other clinical trials or studies.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The effects of probiotics on the postoperative ascending cholangitis | 12 weeks
  To determine the gut microbiota in control of ascending cholangitis before and after pancreaticoduodenectomy through the analysis of microbial community by next generation sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No